CLINICAL TRIAL: NCT01570621
Title: Personalized Peroral Endoscopic Myotomy for Achalasia
Acronym: POEM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zou Xiaoping, vice-principal, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DrumTower206-01
Record Dates: First submitted 2012-04-01; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Achalasia; Postoperative Complications
Keywords: achalasia; peroral endoscopic myotomy; LES pressure; postoperative complication; symptom relief; esophageal barium
MeSH Terms: conditions — Esophageal Achalasia; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: peroral endoscopic myotomy — A 3-cm incision is made into the mucosa after injection of saline and methylene blue. A submucosal tunnel is created from the mid-esophagus to the gastric cardia by a triangle-tip knife. The circular muscle fibers or full-thickness muscle are divided by the triangle-tip knife over a length of 6-20 cm on the esophagus, starting 3 cm below the initial mucosal incision, and extended 3-4cm onto the gastric cardia. The mucosal entry site is closed using standard endoscopic clips at last.

SUMMARY:
Achalasia is a rare esophageal motility disorder, characterized by incomplete lower esophageal sphincter relaxation, increased Lower esophageal sphincter (LES) tone, and aperistalsis of the esophagus. Typical clinical symptoms are dysphagia,regurgitation and chest pain. Traditional treatments include endoscopic balloon dilatation or botulinum toxin injection, laparoscopic Heller myotomy with or without a partial fundoplication. Peroral endoscopic myotomy (POEM) has been developed as a further endoscopic effective and minimal invasive treatment. The aim of this study is to investigate the efficacy and safety of POEM in our department, and to assess short-term and long-term efficacy of POEM by using Stooler score, Echardt score, esophageal barium and manometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as achalasia according to symptoms, esophageal barium,manometry and esophagogastroduodenoscopy
* Age over 18 years old
* Signed written informed consent

Exclusion Criteria:

* Patients with previous surgery of the stomach or esophagus
* With known coagulopathy
* Active esophagitis,eosinophilic esophagitis or Barrett's esophagus
* Pregnancy
* Stricture of the esophagus
* Hiatal hernia > 2cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
symptom relief | 1-12months
  compare patients' symptoms before and after POEM at 1 month, 12 months.
Lower esophageal sphincter pressure | 1-12months
  compare patients's lower esophageal sphincter pressure before and after POEM at 1 month,12 months.
improvement of esophageal barium | 1-12 months
  compare esophageal barium before and after POEM at 1 months,12 months
Postoperative complications | 0-12months
  postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Tingsheng Ling, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937